CLINICAL TRIAL: NCT07053709
Title: Screening for Hyperuricemia in Patients With Metabolic Associated Fatty Liver Disease (MAFLD)
Acronym: SUMA
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohammed Abdel Mowgod, Clinical lecturer, Assiut University
Other Study IDs: 4-2025-300626
Record Dates: First submitted 2025-06-21; First posted 2025-07-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-06

CONDITIONS: Hyperuricemia and MAFLD
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples were collected to assess the following parameters: serum uric acid, liver function tests: albumin, bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transpeptidase (GGT), and alkaline phosphatase (ALP), lipid profile: total cholesterol, triglycerides, and high-density lipoprotein (HDL), complete blood count (CBC): hemoglobin (Hb), white blood cell count (WBC), and platelet count (PLT), viral markers: anti-HCV, HBsAg), plasma high-sensitivity C-reactive, protein, HbA1c.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Due to the established correlation between serum uric acid (SUA) levels and metabolic associated fatty liver disease (MAFLD), this study aims to screen for hyperuricemia in all patients diagnosed with MAFLD.

The ultimate goal is to support the management of MAFLD and improve patients' quality of life by reducing both morbidity and mortality.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) has become increasingly prevalent in recent years and is now considered a leading cause of chronic liver disease worldwide, representing a major global public health challenge.

This growing prevalence is largely attributed to changes in lifestyle and dietary habits, making NAFLD the most common chronic liver condition globally, with an estimated global prevalence of 30.1%.

Recently, an international expert consensus proposed redefining NAFLD as metabolic dysfunction-associated fatty liver disease (MAFLD) to better reflect the disease's underlying metabolic basis. The diagnosis of MAFLD is based on the presence of hepatic steatosis in more than 5% of hepatocytes, in the absence of excessive alcohol intake or other causes of chronic liver disease. The diagnosis also requires at least one of the following three criteria: (1) overweight or obesity, (2) type 2 diabetes mellitus, or (3) evidence of metabolic dysregulation. Metabolic dysregulation is defined by the presence of at least two of the following abnormalities: increased waist circumference, elevated blood pressure, dyslipidemia, prediabetes, insulin resistance, or elevated plasma C-reactive protein (CRP) levels.

"Burned-out" NAFLD has been suggested as a potential hidden cause of cryptogenic cirrhosis. Therefore, early detection and management of NAFLD and its metabolic risk factors are critical to prevent disease progression and hepatic failure.

Uric acid (UA) is the final product of purine metabolism in the liver, with xanthine oxidase (XO) catalyzing the conversion of hypoxanthine to xanthine and subsequently to UA.

Abnormal UA metabolism is associated with various systemic diseases, including hypertension, atherosclerosis, diabetes mellitus, and dyslipidemia.

In recent years, increased interest has been directed toward the relationship between serum uric acid (SUA) levels and NAFLD severity. SUA has been identified as an independent risk factor significantly correlated with NAFLD severity, regardless of other metabolic markers. Studies have shown a 21% increase in NAFLD risk for every 1 mg/dL rise in SUA, and hyperuricemia is associated with a higher risk of advanced liver fibrosis in NAFLD patients.

Given the strong association between SUA levels and NAFLD progression, SUA-lowering therapy has emerged as a potential strategy for improving liver outcomes. Xanthine oxidase inhibitors, such as febuxostat and allopurinol, are commonly used to reduce SUA levels and have shown promise in improving liver histology in patients with NAFLD

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 18 years.
* Diagnosis of MAFLD based on abdominal ultrasonography or other validated imaging techniques.

Exclusion Criteria:

* Patients aged 18 years or younger.
* Pregnant individuals.
* Presence of any malignancy.
* Diagnosis of type 1 diabetes mellitus (T1DM).
* Patients with fatty liver disease who have previously undergone bariatric surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients with metabolic-associated fatty liver disease (MAFLD) were enrolled. Data collected included demographics, clinical history (comorbidities such as diabetes, hyperlipidemia, and hypertension), lifestyle factors (including alcohol intake), anthropometric measures (BMI, waist circumference), blood tests (uric acid, liver enzymes, lipid profile, CBC, HbA1c, hs-CRP, viral markers), and imaging by transient elastography (FibroScan with CAP).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Search for hyperuricemia in every patient with MAFLD | At diagnosis and follow up after 6 month
  1. Prevalence of Hyperuricemia in Patients with MAFLD Description:Number of participants diagnosed with hyperuricemia based on serum uric acid levels.Time Frame:At diagnosis and 6-month follow-up, Unit of Measure:Number of participants
  2. Mean Serum Uric Acid Level Description:Average serum uric acid concentration among study participants. Time Frame:At diagnosis and 6-month follow-up, Unit of Measure:mg/dL
  3. Alanine Aminotransferase (ALT) Level Description:Mean ALT level to assess liver function. Time Frame: At diagnosis and 6-month follow-up. Unit of Measure: IU/L
  4. Aspartate Aminotransferase (AST) Level Description:Mean AST level to assess liver function.Time Frame:At diagnosis and 6-month follow-upUnit of Measure:IU/L
  5. Alkaline Phosphatase (ALP) Level Description:Mean ALP level to assess liver function.Time Frame:At diagnosis and 6-month follow-up. Unit of Measure:IU/L
  6. Serum Albumin Level:Mean serum albumin concentration.Time Frame:At diagnosis and 6-month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Assiut University, Principal Investigator — Assiut University